CLINICAL TRIAL: NCT06315517
Title: A Randomized Controlled Crossover Trial to Assess Tolerance, Gastrointestinal Distress & Preference for Milks Varying in Casein Types & Lactose Content
Brief Title: Double Crossover Casein Type Tolerance Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Andrew Fruge, Associate Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 23-552 MR 2404; 1792-23P (Other Grant/Funding Number: The Dairy Alliance)
Record Dates: First submitted 2024-03-02; First posted 2024-03-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Dairy Intolerance; Healthy Adults
Keywords: A2 casein; A1 casein; fluid milk; lactose; dairy
MeSH Terms: interventions — Milk

STUDY DESIGN:
Intervention Model Description: Randomized controlled, double-blinded, double-crossover trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional lactose-free milk first (Experimental): Participants will consume conventional lactose-free milk first, then each of the other milk types in random order
  Interventions: Other: Conventional lactose-free cow's milk; Other: Nonconventional (A2) cow's milk; Other: Nonconventional (A2) lactose-free cow's milk
- Non-conventional (A2) lactose-free milk first (Experimental): Participants will consume non-conventional (A2) lactose-free milk first, then each of the other milk types in random order
  Interventions: Other: Conventional lactose-free cow's milk; Other: Nonconventional (A2) cow's milk; Other: Nonconventional (A2) lactose-free cow's milk
- Non-conventional (A2) milk first (Experimental): Participants will consume non-conventional (A2) milk first, then each of the other milk types in random order
  Interventions: Other: Conventional lactose-free cow's milk; Other: Nonconventional (A2) cow's milk; Other: Nonconventional (A2) lactose-free cow's milk

INTERVENTIONS:
Other: Conventional lactose-free cow's milk — Participants will receive conventional lactose-free cow's milk as follows:
  On Day 1, participants will receive 50mg casein/kg/bw (~125ml milk). On Day 3, participants will receive 100mg casein/kg/bw (~250ml milk). On Day 5, participants will received 200mg casein/kg/bw (~500ml milk). During test phases, breath hydrogen and methane will be measured every thirty minutes for three hours, and blood glucose will be measured every thirty minutes for two hours. Gastrointestinal symptoms will be assessed with visual analog scales for the following 24 hours. There will be a 7-10 day wash out period in between test phases.
Other: Nonconventional (A2) cow's milk — Participants will receive nonconventional (A2) cow's milk as follows:
  On Day 1, participants will receive 50mg casein/kg/bw (~125ml milk). On Day 3, participants will receive 100mg casein/kg/bw (~250ml milk). On Day 5, participants will received 200mg casein/kg/bw (~500ml milk). During test phases, breath hydrogen and methane will be measured every thirty minutes for three hours, and blood glucose will be measured every thirty minutes for two hours. Gastrointestinal symptoms will be assessed with visual analog scales for the following 24 hours. There will be a 7-10 day wash out period in between test phases.
Other: Nonconventional (A2) lactose-free cow's milk — Participants will receive nonconventional (A2) lactose-free cow's milk as follows:
  On Day 1, participants will receive 50mg casein/kg/bw (~125ml milk). On Day 3, participants will receive 100mg casein/kg/bw (~250ml milk). On Day 5, participants will received 200mg casein/kg/bw (~500ml milk). During test phases, breath hydrogen and methane will be measured every thirty minutes for three hours, and blood glucose will be measured every thirty minutes for two hours. Gastrointestinal symptoms will be assessed with visual analog scales for the following 24 hours. There will be a 7-10 day wash out period in between test phases.

SUMMARY:
The investigators will recruit 45 fluid milk avoiding adults to participate in a five-week double-blind, double-crossover study in which the physiological responses to increasing doses of lactose-free (A1-rich milk), A2 milk, and lactose-free A2 milk will be explored.

DETAILED DESCRIPTION:
Dairy provides essential nutrients and dairy products and are among the best quality and bioavailable protein sources available to humans. Milk protein allergy is extremely rare outside of childhood, and lactose intolerance is highly variable among ethnicities. Nonetheless, many adults avoid fluid milk and dairy products unnecessarily. Recent studies suggest that dairy intolerant individuals are having gastrointestinal reactions specifically to the bioactive metabolites (specifically, beta-casomorphin-7[BCM-7]) of casein protein subtype A1, and consuming milk void of A1 and rich in A2 casein alleviates symptoms.

The investigators will recruit 45 fluid milk avoiding adults to participate in a five-week double-blind, double-crossover study in which physiological responses to increasing doses of lactose-free (A1-rich milk), A2 milk, and lactose-free A2 milk will be explored. Enrollment assessments will include a comprehensive metabolic panel, diet history, and medical history questionnaires. Stool samples will be collected at the beginning and end of each of the 3 test phases (6 total samples per participant). Each test phase will last 6 days long, during which participants will receive increased doses of casein every 2 days.

On Day 1, participants will receive 50mg casein/kg/bw (~125ml milk). On Day 3, participants will receive 100mg casein/kg/bw (~250ml milk). On Day 5, participants will received 200mg casein/kg/bw (~500ml milk). During test phases, breath hydrogen and methane will be measured every thirty minutes for three hours, and blood glucose will be measured every thirty minutes for two hours. Gastrointestinal symptoms will be assessed with visual analog scales for the following 24 hours. There will be a 7-10 day wash out period in between test phases.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18+
* Currently avoid liquid milk
* Can read and speak English

Exclusion Criteria:

* Diagnosis of milk protein allergy
* Diagnosis of Crohn's Disease, Ulcerative Colitis, Celiac Disease, or Peptic Ulcer Disease or Gastroparesis
* Using antibiotic or antiviral medications within 30 days prior to study start
* Undergoing chemotherapy, or using any investigational drugs within 30 days prior to study start
* Pregnant or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Distress Scores | 24 hours after each sample challenge
  Changes in gastrointestinal distress measured via visual analog scales that range from 0 (no symptoms) to 100 cm (severe symptoms). Lower values are optimal.

SECONDARY OUTCOMES:
Breath Hydrogen (ppm) | Three hours after each sample challenge
  Breath hydrogen will be measured via QuinTron BreathTracker SC Analyzer every 30 minutes for three hours beginning immediately prior to each sample challenge. Lower levels are optimal.
Breath Methane (ppm) | Three hours after each sample challenge
  Breath methane will be measured via QuinTron BreathTracker SC Analyzer every 30 minutes for three hours beginning immediately prior to each sample challenge. Lower levels are optimal.
Blood Glucose (mg/dl) | Two hours after each sample challenge
  Capillary finger sticks will determine blood glucose levels for two hours beginning immediately prior to each sample challenge. Minimal deviations from baseline are optimal.
Stool microbiome composition | One week after each sample challenge
  16S changes in microbiome alpha diversity. Higher levels are optimal.
Stool Beta-casomorphin-7 (BCM-7) | One week after each sample challenge
  Fecal samples preserved in aqueous solution will be analyzed for casein metabolite, BCM-7. Lower levels are optimal.
Stool intestinal fatty acid binding protein (I-FABP) | One week after each sample challenge
  Fecal samples preserved in aqueous solution will be analyzed for intestinal permeability marker, I-FABP. Lower levels are optimal.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Frugé, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States